CLINICAL TRIAL: NCT00312364
Title: Safety and Efficacy Study of MRE0094 to Treat Chronic, Neuropathic, Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRE0094P-201
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Foot Ulcer, Diabetic; Diabetes Complications
Keywords: toe ulcer; heel ulcer; foot ulcer; diabetic feet; diabetic foot; complications of diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications; digital ulcers; Foot Ulcer | interventions — 2-(2-(4-chlorophenyl)ethoxy)adenosine

INTERVENTIONS:
Drug: MRE0094

SUMMARY:
This is a clinical research study of an experimental topical drug for the treatment of chronic, neuropathic, diabetic foot ulcers.

Patients participating in the study may receive an active drug (MRE0094), inactive drug (placebo), or a gel used to treat diabetic foot ulcers currently available for sale in the United States. What treatment a patient will receive is determined by chance (like drawing a number from a hat). All patients will receive additional care for diabetic foot ulcers during the study.

Participation in the study can be up to 4½ months.

ELIGIBILITY:
Inclusion Criteria:

Participants included in the study must:

* Have type 1 or type 2 diabetes mellitus.
* Have problems with the nerves in their feet.
* Have an ulcer on the bottom surface of their foot that has been present for 3 weeks or more and is of sufficient size to qualify for the study.
* Be able to apply study drug to their ulcer, or have a caregiver do it.
* Be able to visit the doctor regularly during the 4½ month study.

Exclusion Criteria:

Participants may not participate in the study if:

* Their ulcer is caused by bad blood flow to their foot.
* Their ulcer is infected.
* They cannot wear a special boot during the study to take pressure off the ulcer.
* They have certain other diseases, or are using certain types of drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of complete healing of target ulcer at endpoint or 90 days, whichever is earlier.

SECONDARY OUTCOMES:
Time to closure and percent reduction in surface area of the target ulcer.
Incidence, intensity, and seriousness of adverse events. Changes in irritation scores.

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - Palo Verde Foot and Ankle, Bullhead City, Arizona
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Associated Foot & Ankle Specialists, LLC, Phoenix, Arizona
  - Aung Foot Health Clinics & Advanced Wound Care, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Vertex Clinical Research, Bakersfield, California
  - Roy O. Kroeker, DPM, Fresno, California
  - Innovative Medical Technologies, Los Angeles, California
  - UCSD Wound Treatment and Research Center, San Diego, California
  - Bay Area Foot Care, San Francisco, California
  - Walter F. D'Costa, DPM, Santa Rosa, California
  - Diabetic Foot & Wound Center, Denver, Colorado
  - North American Center for Limb Preservation, New Haven, Connecticut
  - Christiana Care Health Systems Wound Care Center, Wilmington, Delaware
  - Countryside Foot and Ankle Center, Clearwater, Florida
  - Karr Foot & Leg Centers, Lakeland, Florida
  - University of Miami, Miami, Florida
  - Baptist Hospital, Pensacola, Florida
  - Doctor's Research Network, South Miami, Florida
  - Dr. Robert J. Snyder, Tamarac, Florida
  - Ankle and Foot Specialist of Atlanta, Lithonia, Georgia
  - Podiatry Center of Idaho, PLLC, Boise, Idaho
  - Adam S. Landsman, DPM, PhD, FACFAS, Highland Park, Illinois
  - Advocate Lutheran General Hospital, Niles, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Thomas Kevin Brattain, DPM, Peoria, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Welborn Clinic, Evansville, Indiana
  - The Wound Healing Center, Terre Haute, Indiana
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - David Fivenson, MD, Dermatology, PLLC, Ann Arbor, Michigan
  - Foot Healthcare Associates, Livonia, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Foot & Ankle Physicians, Union, New Jersey
  - St. John's Queens Hospital, Elmhurst, New York
  - North Shore Podiatry Group, Port Jefferson Station, New York
  - Calvary Hospital, The Bronx, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - UNC Wound Care Clinic, Durham, North Carolina
  - Eastern Carolina Foot & Ankle Specialists, Greenville, North Carolina
  - Bone, Spine, Sports Center, Bismarck, North Dakota
  - Austintown Podiatry Associates, Inc., Austintown, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Optimed Research, LLC, Columbus, Ohio
  - Lehigh Valley Podiatry Associates, Allentown, Pennsylvania
  - Advanced Regional Center for Ankle and Foot Care, Altoona, Pennsylvania
  - UPMC Horizon, Farrell, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Foot and Ankle Institute, Philadelphia, Pennsylvania
  - Prigoff-Bowers, LLP, Dallas, Texas
  - Limb Salvage Center, Dallas, Texas
  - South Texas Foot Institute, Floresville, Texas
  - Memorial Hermann Wound Center, Houston, Texas
  - Southwest Regional Wound Care Center, Lubbock, Texas
  - Barrett Quality Medical Interests, LP, San Antonio, Texas
  - San Antonio Podiatry Associates, PC, San Antonio, Texas
  - Richard G. Seegmiller, DPM, Bountiful, Utah
  - Douglas C. Flegal, DMP, FACFAS, Salt Lake City, Utah
  - Atlantic Foot & Ankle Center, Virginia Beach, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin